CLINICAL TRIAL: NCT05594940
Title: Heart Failure Monitoring With a Portable Ultrasound Device With Artificial Intelligence Assisted Tools: A Multi-Phase Observational Feasibility Study
Status: Terminated | Type: Observational
Why Stopped: Data Analysis
Sponsor: Butterfly Network (Industry)
Responsible Party: Sponsor
Other Study IDs: BN03
Record Dates: First submitted 2022-10-20; First posted 2022-10-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Congestive Heart Failure
Keywords: CardioMEMS; iQ+; Home; CHF; B-Lines
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
The primary objective of this study is to evaluate the feasibility of a novel app to facilitate heart failure patients to acquire lung ultrasound images and evaluate the quality of those images to expert scans, and to evaluate for relationships between the ultrasound data and pulmonary pressure data from the Abbott CardioMEMS system.

DETAILED DESCRIPTION:
Feasibility study to compare an investigational Artificial Intelligence (AI) Auto B-line tool measurement on Lung Ultrasound (US) images acquired with an AI assisted guidance tool by novice ultrasound clinicians and heart failure (HF) patients, to standard of care heart failure monitoring of pulmonary artery pressure measured by the Abbott CardioMEMS system.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of heart failure at least three months prior to the date of consent
2. HF currently managed with the Abbott CardioMEMS device
3. Able to read and write in English.
4. At least 18 years of age or older on the date of consent.
5. Willing and able to provide written consent to participation
6. Expressed willingness to capture AI assisted US recordings immediately before or after taking their CardioMEMS measurements
7. Access to WiFi or cellular data connection at home
8. In the opinion of the investigator or delegate the subject, must be capable of complying with study procedures.

Exclusion Criteria:

1. Previous experience using an ultrasound device on themselves or others
2. Women who are pregnant or plan to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CHF patients with CardioMEMS devices
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Patients Image Quality | Study Completion (91 days)
  Image quality comparisons between ultrasound scans performed by heart failure patients using the study app to traditional ultrasound scans performed by trained clinicians
Novice Image Quality | Study Completion (91 days)
  Image quality comparisons between ultrasound scans performed by novice clinicians using the study app to traditional ultrasound scans performed by trained clinicians
B-Line count CardioMEMS comparison | Study Completion (91 days)
  Relationship comparisons between ultrasound data from exams performed by heart failure patients using the study app (both in clinic and at home) and ultrasound exams performed by novice clinicians to pulmonary pressure data from the Abbott CardioMEMS system

SECONDARY OUTCOMES:
Ease of use | Study Completion (91 days)
  Patient and novice clinician reported ease of use and satisfaction based on responses to user surveys.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - John Muir Health Hospital, Concord Medical Center, Concord, California
  - John Muir Health Hospital, Walnut Creet Medical Center, Walnut Creek, California

IPD SHARING:
Plan to Share IPD: No